CLINICAL TRIAL: NCT00869102
Title: Characterization of Beta Cell Failure
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Hans-Ulrich Haering, UIniversity of Tübingen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: BET-001
Record Dates: First submitted 2009-03-23; First posted 2009-03-25 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2009-03

CONDITIONS: Diabetes; Metabolic Syndrome
Keywords: IGT; IFG
MeSH Terms: conditions — Diabetes Mellitus; Metabolic Syndrome | interventions — Glucagon-Like Peptide 1

ARMS (1):
- GLP-1 (Experimental)
  Interventions: Drug: GLP-1

INTERVENTIONS:
Drug: GLP-1 — intravenous, 124,5 pmol/kg body weight

SUMMARY:
The purpose of this study is to characterise beta cell function in subjects who despite taking part in a diabetes prevention program (life style intervention with diet and exercise) exhibit impaired glucose tolerance and beta cell dysfunction.

DETAILED DESCRIPTION:
We have identified a subgroup of individuals with a good compliance to lifestyle intervention to prevent diabetes who lose body weight and increase insulin sensitivity, however they remain impaired glucose tolerant. These individuals show a deterioration in insulin secretory function.

We will identify a highly selected group of subjects with prediabetes that displays a large defect in insulin secretory function.We will study 50 individuals who display these characteristics and 50 subjects who do not display these characteristics. Their insulin secretion capacity in response to different secretagogues (glucose, GLP-1, arginine) will be studied. We expect to detect new pathophysiologic aspects that lead to beta cell failure particularly in this group.

ELIGIBILITY:
Inclusion Criteria:

* Impaired glucose tolerance
* BMI 16-40 kg/m²

Exclusion Criteria:

* chronic disease
* anemia
* therapy with insulin or cortisone

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-05; Primary Completion 2010-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Insulin secretion | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- University of Tübingen, Tübingen, Germany